CLINICAL TRIAL: NCT02179970
Title: To Assess the Safety of Continuous IV Administration of the CXCR4 Antagonist, Plerixafor (Mozobil), and Assess Its Impact on the Immune Microenvironment in Patients With Advanced Pancreatic, High Grade Serous Ovarian and Colorectal Adenocarcinomas.
Brief Title: To Assess the Safety of Continuous IV Administration of Plerixafor in Patients With Advanced Pancreatic, Ovarian and Colorectal Cancers
Acronym: CAM-PLEX
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CCTU- Cancer Theme (Other)
Collaborators: Sanofi (Industry); Stand Up To Cancer (Other); CRUK Cambridge Institute (Unknown); Lustgarten Foundation (Other); National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor-Investigator, CCTU- Cancer Theme, Professor Duncan Jodrell, Cambridge University Hospitals NHS Foundation Trust
Organization: Cambridge University Hospitals NHS Foundation Trust (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAM-PLEX; 2014-000117-31 (EudraCT Number)
Record Dates: First submitted 2014-07-01; First posted 2014-07-02 (Estimated); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Pancreatic Adenocarcinoma Metastatic; Ovarian Serous Adenocarcinoma; Colorectal Cancer Metastatic
Keywords: Advanced pancreatic cancer; Advanced ovarian cancer; Advanced colorectal cancer; Metastatic pancreatic cancer; Metastatic ovarian cancer; Metastatic colorectal cancer
MeSH Terms: conditions — Pancreatic Neoplasms; Ovarian Neoplasms; Colorectal Neoplasms | interventions — plerixafor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Plerixafor (Mozobil) (Other): Plerixafor (Mozobil), continuous 7 day IV infusion. Starting at a dose of 20 ug/kg/hr, and subsequent dose levels of 40, 80 and 120 ug/kg/hr.
  Interventions: Drug: Plerixafor

INTERVENTIONS:
Drug: Plerixafor — A continuous 7 day intravenous infusion, starting at a dose of 20 ug/kg/hr, and subsequent dose levels of 40, 80 and 120 ug/kg/hr.
  Other Names: Mozobil

SUMMARY:
Pancreatic, ovarian and colorectal cancers are difficult to treat using chemotherapy and immune therapies.Currently most patients are offered treatment with a standard chemotherapy drug depending on their cancer type. Recently, laboratory studies have shown that a drug called plerixafor may help the body to overcome resistance to immune therapy.

The purpose of this study is to find out if the study drug has the same effect on patients with advanced pancreatic, ovarian or colorectal cancer, as we have seen in our laboratory experiments, and find out the right dose of the study drug to give. This is a 'dose escalation study'. Patients will be recruited slowly and the study team will closely monitor the effect the drug has, until they find the best dose to give. As part of this study, blood and tumour samples will be collected and analysed in our laboratories and the patients cancer will be monitored using two imaging techniques, CT and FDG-PET scans.

DETAILED DESCRIPTION:
This is a prospective, non-randomised, open label, Phase I, dose escalation study of plerixafor (MozobilTM) in patients with histological documentation of advanced pancreatic, high grade serous ovarian or colorectal adenocarcinoma. We will investigate the feasibility of administering plerixafor in terms of safety, and will try to identify the proof of mechanism in patients.

This study is required to establish whether relevant plasma concentrations of plerixafor can be achieved safely in patients with advanced pancreatic, high grade serous ovarian and colorectal cancer.

Plerixafor (Mozobil) will be administered as a continuous 7 day intravenous infusion, starting at a dose of 20 ug/kg/hr, and subsequent dose levels of 40, 80 and 120 ug/kg/hr (as an inpatient for at least the initial 48 hours). 3 patients will be entered sequentially (at least 1 week apart), using a standard 3+3, Phase I trial design. Up to 28 patients will be recruited.

ELIGIBILITY:
Inclusion Criteria:

* Aged 16 years or over at the time of signing informed consent form.
* Dose escalation phase only: Patients with inoperable, histologically proven locally advanced or metastatic pancreatic, high grade serous ovarian or colorectal adenocarcinoma, refractory to conventional chemotherapy or a patient who has declined conventional chemotherapy. OR;
* Expansion phase only: Patients with inoperable, histologically proven locally advanced or metastatic pancreatic, refractory to conventional chemotherapy or a patient who has declined conventional chemotherapy.
* Tumour lesions considered to be accessible for core biopsy and immunostaining assessment.
* ECOG performance status 0-1.
* Life expectancy of at least 12 weeks.
* All women of child-bearing potential and all sexually active male patients must agree to use effective contraception methods throughout the study and for 3 months after the final dose of study drug.

Exclusion Criteria:

* Inadequate haematological function defined by:
* Absolute neutrophil count (ANC) <1.5 x 109/L
* Absolute lymphocyte count < normal level for institution
* Haemoglobin <9.0 g/dL (90 g/L) (may be increased to this level with transfusion as long as there is no evidence of active bleeding)
* Platelets <100 x 109/L
* Clotting; INR >1.3
* Inadequate renal function defined by calculated creatinine clearance by Cockcroft-Gault of <50 ml/min.
* Inadequate hepatic function defined by:
* Aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) >2.5 x upper limit of normal (ULN) or >5 x in the presence of liver metastases
* Total bilirubin >1.5 x ULN
* Current treatment (within 28 days of entry) with chemotherapy, steroids or other immunosuppressive drugs.
* Significant acute or chronic medical or psychiatric condition, disease or laboratory abnormality which in the judgment of the Investigator would place the patient at undue risk or interfere with the study.
* Cardiac co-morbidity:
* Past history of significant rhythm disturbance (e.g. SVT, AF or ventricular irregularities)
* Requirement for pacemaker.
* Myocardial infarction in the previous 6 months.
* Known medical history of proven postural hypotension.
* Active infection.
* Patients with known allergy to plerixafor or its excipients.
* Patients known to have hepatitis B, hepatitis C or HIV infection.
* Women, who are pregnant, plan to become pregnant or are lactating (during the study or for up to 3 months after the last dose)

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2018-12-14 (Actual); Study Completion 2018-12-14 (Actual)

PRIMARY OUTCOMES:
Safety of Investigational Medicinal Product (IMP) | 24 months
  Determining the causality of adverse events (AEs) and serious adverse events (SAEs)

SECONDARY OUTCOMES:
Pharmacokinetics of the Investigational Medicinal Product (IMP) within the body. | 24 months
  Determining the absorption, distribution, metabolism, and excretion rates of the IMP through concentration rates in plasma samples.

OTHER OUTCOMES:
Disease status | 24 months
  Anticancer impact following treatment with plerixafor.
Disease status | 24 months
  Metabolic tumour changes using FDG-PET.

CONTACTS AND LOCATIONS:
Overall Officials: Professor Duncan Jodrell, Study Director — CRUK Cambridge Institute and the University of Cambridge
Locations (1):
- Addenbrookes Hospital, Cambridge, United Kingdom

REFERENCES:
- See also: Cambridge Pancreatic Centre, University of Cambridge — http://www.cambridge-pcc.org/